CLINICAL TRIAL: NCT01598168
Title: Rivaroxaban for Treatment of Patients With Suspected or Confirmed Heparin-Induced Thrombocytopenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-02-09
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Heparin-induced Thrombocytopenia
Keywords: rivaroxaban; treatment; venous thromboembolism; arterial thromboembolism; thrombocytopenia
MeSH Terms: conditions — Venous Thromboembolism; Thrombocytopenia | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rivaroxaban (Experimental): Rivaroxaban 15 mg bid until HIT excluded by local laboratory assay or platelets recovered. If HIT positive and platelets have recovered, patients will receive rivaroxaban 20 mg od until Day 30.
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 15 mg bid until HIT excluded by local laboratory assay or platelets recovered. If HIT positive and platelets have recovered, patients will receive rivaroxaban 20 mg od until Day 30.
  Other Names: Xarelto

SUMMARY:
Heparin is an anticoagulant (blood thinner) that is commonly used to treat patients with heart attacks and patients with blood clots in their legs or lungs (venous thrombosis). Some patients develop an allergic reaction to heparin, a condition called heparin-induced thrombocytopenia (HIT). HIT makes blood clot, which is the opposite of what heparin was designed to do. These blood clots can lead to heart attacks, strokes, limb amputations, and death. The objective of this 200 patient study is to determine if a new blood thinner called rivaroxaban (Xarelto) can be used to treat HIT. Rivaroxaban can be taken by mouth, does not require blood testing, and had a low risk of bleeding when it was used to treat blood clots in other clinical trials. If this study shows that rivaroxaban can be used to treat HIT, there will be two very important benefits. For patients with HIT, the benefit will be having a safe, and easy-to-use drug to protect them from developing further life or limb-threatening blood clots. For the Canadian health care system, the benefit will be having a drug that is much less expensive than the drugs currently used to treat HIT.

DETAILED DESCRIPTION:
Consecutive adult patients with an intermediate or high clinical probability for HIT (according to the clinical prediction rule called the "4T's Score) will receive rivaroxaban 15 mg bid while awaiting confirmation or exclusion of HIT by the local laboratory assay. Patients who are confirmed to have HIT by the local laboratory assay will continue to receive rivaroxaban 15 mg bid until their platelet count ≥ 150 or until end of study (Day 30). At the time of platelet count recovery (typically 4-7 days), they will be transitioned to a maintenance dose of rivaroxaban (20 mg od) for a maximum of 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with 4T's Score greater than or equal to 4.

Exclusion Criteria:

* Require ongoing anticoagulant therapy for a mechanical heart valve.
* Severe renal insufficiency (CrCl<30 ml/min)
* Hepatic disease (including Child-Pugh B and C) associated with coagulopathy and a clinically relevant bleeding risk
* Inability to take oral medications.
* Ongoing requirement for systemic treatment with azole-antimycotics (except fluconazole) or HIV-protease inhibitors or strong CYP3A4 inducers
* Clinically significant active bleeding or lesions at increased risk for bleeding within the last 6 months
* Platelet count less than 80 and an ongoing need for antiplatelet therapy may be excluded at the discretion of the investigator
* Pregnant or a woman of child-bearing potential not using an adequate birth control method
* Hypersensitivity to rivaroxaban or to any ingredient in the formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Incidence of new symptomatic venous and arterial thromboembolism in the study population. | 30 days

SECONDARY OUTCOMES:
Incidence of symptomatic venous and arterial thromboembolism and major bleeding in patients while on-treatment with rivaroxaban. | 30 days
Duration of time to platelet recovery in patients with Serotonin Release Assay (SRA) confirmed HIT | 30 days
Incidence of venous and arterial thromboembolism in patients with SRA confirmed HIT who receive rivaroxaban. | 30 days
Major bleeding in the entire study population and in patients with SRA confirmed HIT who receive rivaroxaban. | 30 days
To collect data to prospectively validate a new clinical prediction rule for HIT | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Lori-Ann Linkins, MD, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences - Juravinski Site, Hamilton, Ontario, Canada